CLINICAL TRIAL: NCT04077255
Title: Anti-EGFR Antibody (GC-1118) in Combination With Weekly Paclitaxel as a Second-line Therapy for Gastric and Gastroesophageal Junction Adenocarcinomas With Amplifications
Brief Title: EGFR-targeted Therapy for Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Hark Kyun Kim, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31973
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Adenocarcinoma of the Stomach
Keywords: EGFR
MeSH Terms: interventions — GC1118

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-EGFR (Experimental): Participants will receive GC-1118 in combination with weekly paclitaxel.
  Interventions: Drug: Anti-EGFR antibody in combination with weekly paclitaxel

INTERVENTIONS:
Drug: Anti-EGFR antibody in combination with weekly paclitaxel — Intravenous GC-1118 in combination with weekly paclitaxel for EGFR-amplified cancer cancers as a second-line therapy
  Other Names: GC-1118 in combination with weekly paclitaxel

SUMMARY:
Based on targeted NGS panel results, metastatic gastric cancer patients with gene amplifications will receive either anti-EGFR antibody (GC-1118) in combination with weekly paclitaxel as a second-line therapy.

DETAILED DESCRIPTION:
Participants will receive each treatment if the gastric cancer tissue sample reveals either EGFR gene amplification or strong (3+ or 2+) EGFR immunostaining

ELIGIBILITY:
Key inclusion criteria

1. Histologically-proven gastric and gastroesophageal junction adenocarcinoma
2. Refractory to first-line chemotherapy for metastatic disease
3. Presence of at least 1 measurable lesion according to RECIST version 1.1
4. EGFR gene amplification or strong (3+ or 2+) EGFR immunostaining

Key exclusion criteria

1.Prior exposure to taxane or EGFR-targeted therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | Response rate will be assessed at 8 weeks.
  Response rate will be assessed using CT/MRI according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival | From date of enrollment until the date of first documented progression or the date of death from any cause, whichever came first, will be assessed up to 1 year.
  Time from date of enrollment until the date of first documented progression or the date of death from any cause, whichever came first, will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hark K Kim, M.D.,Ph.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No